CLINICAL TRIAL: NCT05247606
Title: Impact of a Mobile Health Application in Improving Lifestyle and Therapeutic Adherence in Coronary Heart Disease: Randomized Clinical Trial
Brief Title: Impact of Mobile Health in Improving Lifestyle and Therapeutic Adherence in Coronary Heart Disease
Acronym: eMOTIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI-0014-2019
Record Dates: First submitted 2022-02-03; First posted 2022-02-21 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Coronary Disease
Keywords: Coronary Disease; Mobile application; Lifestyle; Clinical trial
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Mobile application
  Interventions: Device: Mobile application
- Control group (No Intervention): Usual care

INTERVENTIONS:
Device: Mobile application — Lifestyle intervention through web-based mobile application
  Arms: Intervention group

SUMMARY:
Cardiovascular diseases are the leading cause of death worldwide. In high-income countries, approximately seventy percent of cardiovascular diseases cases are attributable to modifiable risk factors, with metabolic risk factors (obesity, cholesterol) and tobacco use being the most closely associated.

Secondary prevention of coronary disease is considered essential, since it has contributed significantly to the reduction of morbidity and mortality, by facilitating the adoption and adherence to healthy behaviors, promoting an active lifestyle, and increasing adherence to pharmacological treatment.

Information and communication technologies have been increasingly incorporated into health care systems, including the innovative provision of Cardiac Rehabilitation through a mobile phone or m-health interventions. M-health technology can provide evidence-based guidance in an interactive format that is attractive, easy to use, and reduces healthcare costs.

The objective of this study is to evaluate, through a randomized controlled clinical trial, the effect of an intervention based on a web application of health, mobile Health, on lifestyle (diet, physical activity, and nicotine dependence) and therapeutic adherence in people with coronary heart disease.

The sample will consist of 200 participants, 100 in the intervention group and 100 in the usual care group that will be evaluated at the beginning and 3, 6, and 12 months after hospital discharge regarding sociodemographic, clinical, cardiovascular risk factors, lifestyle, and therapeutic adherence characteristics. The educational intervention, monitoring, and self-monitoring will be carried out using a web-based m-Health tool, mobile phone application. The quantitative primary results will be compared between the two groups using analysis of covariance, adjusting for age and sex. Multivariate analysis will be carried out to examine the association of the intervention with life habits, control of cardiovascular risk factors as well as the evolution after discharge in respect of cardiovascular events, emergency and re-entry views.

DETAILED DESCRIPTION:
Design: A randomized single-blind, parallel-group, controlled clinical trial performed on patients with coronary heart disease who underwent a percutaneous coronary intervention with stent placement in the Cardiology Service of a public reference hospital complex providing specialist care in the province of Cadiz, Spain, in which 1500 coronary interventions procedures are performed per year.

Randomization and Blinding: The randomization and allocation to each group (1:1, intervention and usual care) are based on computer-generated random numbers. The researchers responsible for the study do not participate in the allocation of the participants. Due to the kind of intervention, blinding is not possible when the participants are allocated to groups. To minimize any bias, objective clinical variables are measured in the evaluation visit and the analyses are performed by blinded researchers.

Study Sample: The participants are eligible to participate if they have a confirmed diagnosis of coronary heart disease and undergo percutaneous coronary intervention. Furthermore, the participants must comply with the criteria explained in the section.

Sample Size: To detect a medium effect size of Cohen's d of 0.5 regarding adherence to the Mediterranean diet (8.6 ± 2.0 points), physical activity (216 ±92 minutes/day), nicotine dependence (1.50± 2.14 points), and therapeutic adherence (6.47±1.23 points), a 95% confidence interval and a power of 80%, the sample size is estimated at 80 patients in each group. Assuming a 20% loss to follow-up, 200 participants will be recruited, 100 in each arm, intervention and usual care.

Recruitment: After the percutaneous coronary intervention and during admission, the nurse will recruit eligible patients and their care partners, will ask them to sign the informed consent, perform the initial assessment and organize a programmed visit after 3,6 and 12 months. A card will be provided with the dates of the appointments and a telephone number for any changes.

The participants allocated to the usual care group receive the standard prescribed care and advice about medication, and lifestyle.

Both groups will be provided with written recommendations and an explanation about the standard Mediterranean diet, physical activity, stopping smoking and treatment adherence.

Before hospital discharge, all the patients will be encouraged to follow a healthy lifestyle. Stages of change strategies will be used in addition to a motivational and behavior changing interview. Written information will be provided about risk factors, lifestyle goals, a suggested healthy menu, recommendations about the daily intake of food groups, and the other behavior that the intervention is targeting.

Intervention: The intervention begins during the patient's stay in hospital immediately after a coronary event. The participants from the intervention group and their partner/carer will complete a short online tutorial describing the mobile application accessed using a mobile telephone or tablet. They will be advised to use the application for at least 15 min per day. This time has been considered sufficient for the daily recording of data in the pilot study. The intervention and follow-up will last 12 months. If the patient does not record data for a week, he/she receives a message through the app encouraging him to use it. The patients may resolve any queries using the application's built-in messaging function, to which the nurse will reply through this messaging service or with a telephone call. This avoids many patient visits to the doctor for consultations and reduces human resource needs.

Before the trial, a pilot study was performed with 20 participants to test the application and make any necessary adjustments.

Technical Data of the Website and Application: The responsive online application (user registration, data management, downloading records) is managed via the project website, which acts as an access platform after validation with a password. The web environment enables the application to be executed using any browser. Operating environment: it is an application with remote access to a My Structured Query Language (MySQL) database. Technology development: (a) uses Personal Home Page (PHP ) scripting language ; (b) Asynchronous JavaScript and XML (AJAX) web development techniques. The application runs in the user's browser while it communicates with the server in the background; and (c) Bootstrap open-source tools for designing websites and online applications. Data storage: MySQL database is fast enough to deploy web applications. Data protection: in addition to on-demand backups performed by the software, the web server performs daily backups of all the files, so the data and program are doubly protected. Access privacy: The data are not stored in a local computer but on a web server, meaning they can only be accessed with a password. This web server works with anonymous data and is located in the country to comply with the regulations for the protection of high-level data.

Application Contents: The application has educational texts and videos on healthy lifestyle and therapeutic adherence and allows users to set goals and monitor their food consumption, physical exercise, blood pressure, tobacco use, and compliance with their treatment. It is based on the phases of change theory (attention, retention, memory, action, and motivation), and on making the process pleasing. The user's attention is caught through warnings and bright, attractive colors on the user interface; retention is encouraged by reminders, repetition, and graphs; action is prompted by instructions, advice, and feedback; and motivation to change is boosted by internal comparisons (progress graphs), setting goals, self-monitoring, and feedback. Through its different components participants are encouraged to (1) follow a healthy eating pattern based on the Mediterranean diet aligned with national dietary guidelines; (2) perform a physical activity of duration and intensity in line with the recommendations of their cardiologist; (3) stop smoking; (4) monitor their blood pressure; (5) adhere to their treatment by associating taking medication with daily activities, establishing set times for taking it and with support from a relative, etc.

Components of the Application: A) Provide information encouraging a healthy lifestyle. Through the website, the participants will have access to information on their screens that they can print to help them plan a healthier lifestyle and adhere to their treatment. The application also has a training section for the patient with videos and information about the recommended therapeutic objectives in the clinical practice guidelines regarding food, physical activity, body weight, blood pressure, blood sugar, stopping smoking and adhering to treatment.

B) Self-monitoring. The application has a recording and self-checking function to help patients to self-monitor the skills for each behavioral goal about nutrition, physical activity, tobacco consumption, blood pressure, body weight, capillary blood glucose in patients with diabetes mellitus and treatment adherence.

Training: Session about the Application for patient and carer. The nurse will install the shortcut to the application on the screen of the participant's mobile phone and will record the prescribed treatment including the name, dose, and timetable in the application. The nurse will update the prescription in the application if the doctor changes the treatment. During the training session, the participants learn to use the functions of the application: confirm when medication is taken, record the food consumed and physical activity performed (daily), blood pressure, weight, and tobacco consumption (weekly), and capillary blood glucose in participants with diabetes mellitus (twice a week). The participants can follow their evolution and progress through the graphics generated with the information they have recorded over the previous weeks.

Ethical Considerations:The study will be conducted in agreement with the guidelines and protocols established in the Helsinki Declaration as revised in Fortaleza (Brazil) in October 2013, and complies with Law 14/2007 on Biomedical Research and with European Data Protection Regulations. The Biomedical Research Ethics Committee of the Costa del Sol, Andalusian, approved the project with the reference: 002_jun20_PI-RECAMAR-19. The informed written consent of all the patients will be requested. The application guarantees the security measures regarding the current General Data Protection Regulations in Europe. It also includes data encryption mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Participants with coronary heart disease
* Under the age of 75
* Have a mobile phone, with the ability to receive text messages and with internet access

Exclusion Criteria:

* Severe heart failure
* Physical disability
* Dementia
* Congenital heart disease
* Rheumatic etiology disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Adherence to the Mediterranean diet | Month 3, 6 and 12
  A 14-item Questionnaire of Mediterranean diet adherence (unit of measure: points. Each item is scored 0 or 1. The total Mediterranean diet score ranges from 0 to 14 points. The higher the score, the higher the degree of adherence to the Mediterranean Diet.
Change in Frequency of food consumption | Month 3, 6 and 12
  A Food-frequency questionnaire with 20 food items (unit of measure: number of times per month, week and day
Change in Level of physical activity | Month 3, 6 and 12
  International Physical Activity Questionnaire (IPAQ) (unit of measure: minutes of exercise/ day. Minimum: Walk at least 30 minutes a day, 5 times a week (150 minutes a week). Do higher values represent a better outcome.
Change in Test for nicotine dependence | Month 3, 6 and 12
  (Unit of measure: points. Less than 4 points, low dependency; between 4 and 6 points, medium dependency; equal to or greater than 7 points, high dependency).
Change in Therapeutic adherence | Month 3, 6 and 12
  A 8 items questionnaire (Total score: 8 points. Good therapeutic adherence= 8 points. Poor therapeutic adherence= 1-7 points)
Change in Knowledge about cardiovascular disease using a questionnaire | Month 3, 6 and 12
  A 24-item questionnaire (scale 0-5 each item. Do higher values represent a better outcome)
Change in Usability and satisfaction with the application | Month 3, 6 and 12
  A 22 item questionnaire 22 item questionnaire to assess user acceptability of mobile health interventions. (6-point scale, level of disagreement to agreement with each item concerning the usability of the apps. Do higher values represent a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: MJ Santi, MD, Principal Investigator — University of Cadiz
Locations (1):
- Hospital Puerta del Mar, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cruz-Cobo C, Bernal-Jimenez MA, Calle G, Gheorghe LL, Gutierrez-Barrios A, Canadas D, Tur JA, Vazquez-Garcia R, Santi-Cano MJ. Efficacy of a Mobile Health App (eMOTIVA) Regarding Compliance With Cardiac Rehabilitation Guidelines in Patients With Coronary Artery Disease: Randomized Controlled Clinical Trial. JMIR Mhealth Uhealth. 2024 Jul 25;12:e55421. doi: 10.2196/55421. PMID 39052330
- [Derived] Cruz-Cobo C, Bernal-Jimenez MA, Calle-Perez G, Gheorghe L, Gutierrez-Barrios A, Canadas-Pruano D, Rodriguez-Martin A, Tur JA, Vazquez-Garcia R, Santi-Cano MJ. Impact of mHealth application on adherence to cardiac rehabilitation guidelines after a coronary event: Randomised controlled clinical trial protocol. Digit Health. 2024 Mar 19;10:20552076241234474. doi: 10.1177/20552076241234474. eCollection 2024 Jan-Dec. PMID 38510574